CLINICAL TRIAL: NCT04477993
Title: Randomized, Double-Blind Clinical Trial of Ruxolitinib in Patients With Acute Respiratory Disorder Syndrome Due to SARS-CoV-2 Infection
Brief Title: Ruxolitinib for Acute Respiratory Disorder Syndrome Due to COVID-19
Acronym: RUXO-COVID
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Vanderson Geraldo Rocha (Other)
Responsible Party: Sponsor-Investigator, Vanderson Geraldo Rocha, Full Professor, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32894720.3.0000.0068
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2; SARS-CoV2
Keywords: SARS-CoV2; Severe Acute Respiratory Syndrome Coronavirus 2; Janus Kinase Inhibitors; Safety; Clinical Efficacy; Clinical Trial
MeSH Terms: interventions — Janus Kinase Inhibitors; ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - ruxolitinib (Experimental): Ruxolitinib 5 mg PO b.i.d. for 14 days
  Interventions: Drug: Janus Kinase Inhibitor (ruxolitinib)
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Janus Kinase Inhibitor (ruxolitinib) — 5 mg P.O. b.i.d. for 14 days. Dose reduction will occur if neutrophils < 500/mm3 or platelets <50,000/mm3.
  Arms: Experimental Group - ruxolitinib
Other: Placebo — Placebo tablets P.O. b.i.d. for 14 days.
  Arms: Placebo Group

SUMMARY:
The COVID-19 pandemic has had a dramatic effect in public health worldwide. In Brazil, there have been more than 2 million confirmed cases and over 75,000 deaths since February 26, 2020. Based on reports of a hyperinflammatory state associated with COVID-19, the use of immunosuppressive drugs may be efficacious in the treatment of this disease. JAK inhibitors have been shown to harness inflammation in a number of different pathologic conditions. The aim of the present study is to evaluate the efficacy and safety of JAK inhibitor ruxolitinib in patients with acute respiratory distress syndrome due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with SARS-CoV-2 pneumonia confirmed by RT-PCR or serology (IgA);
* PaO2/FiO2 < 300 (not fully explained by heart failure or volume overload) or SpO2 < 90% on room air.

Exclusion Criteria:

* Symptom onset > 14 days;
* Neutrophil count < 1,000/mm3;
* Platelets < 50,000/mm3;
* ICU care at enrollment;
* On invasive mechanical ventilation at enrollment;
* Current use of experimental therapy for COVID-19 (except: azithromycin or corticosteroids)
* Uncontrolled arterial hypertension;
* Current or previous use of systemic immunosuppressive therapy in the last 30 days;
* Pregnancy or lactation;
* Estimated creatinine clearance < 30 mL/min or receiving CRRT or intermittent hemodialysis;
* Allergy to ruxolitinib;
* Active tuberculosis;
* HIV seropositivity;
* Prior history of progressive multifocal leukoencephalopathy;
* Use of any JAK inhibitor in the last 30 days before study enrollment;
* Not qualifying according to investigators' perception.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
A composite outcome of death or ICU admission or mechanical ventilation at day 14. | 14 days

SECONDARY OUTCOMES:
A composite outcome of death or ICU admission or mechanical ventilation at day 28 | 28 days
Time to treatment failure | 28 days
  ICU admission, mechanical ventilation, death or consent withdrawal
Overall survival at days 14 and 28 | 14 and 28 days
Cumulative incidence of ICU admission rate at days 14 and 28 | 14 and 28 days
Cumulative incidence of mechanical ventilation at days 14 and 28 | 14 and 28 days
Duration of hospital stay | 28 days
Duration of ICU stay | 28 days
Duration of mechanical ventilation | 28 days
Duration of non-invasive ventilation | 28 days
Secondary hemophagocytic syndrome rate | 28 days
Cumulative incidence nosocomial infection rate at days 14 and 28 | 14 and 28 days
Incidence of discontinuation of oxygen supplementation at days 14 and 28 | 14 and 28 days
Rate of grade 1-2 and 3-5 emerging adverse events at day 28 | 28 days
Cumulative dose of methylprednisolone at days 14 and 28 | 14 and 28 days
Change in PaO2/FiO2 ratio from baseline to days 14 and 28 | 14 and 28 days
Change in interleukin 6 levels [pg/mL] from baseline to days 14 and 28 | 14 and 28 days
Change in d-dimer levels [ng/mL] from baseline to days 14 and 28 | 14 and 28 days
Change in fibrinogen levels [mg/dL] from baseline to days 14 and 28 | 14 and 28 days
Change in ferritin levels [ng/mL] from baseline to days 14 and 28 | 14 and 28 days
Change in C reactive protein levels [mg/L] from baseline to days 14 and 28 | 14 and 28 days
Change in alanine aminotransferase [U/L] from baseline to days 14 and 28 | 14 and 28 days
Change in aspartate aminotransferase [U/L] from baseline to days 14 and 28 | 14 and 28 days
Change in creatinine levels [mg/dL] from baseline to days 14 and 28 | 14 and 28 days
Change in glucose levels [mg/dL] from baseline to days 14 and 28 | 14 and 28 days
Change in hemoglobin levels [g/dL] from baseline to days 14 and 28 | 14 and 28 days
Change in platelet count [x10ˆ3/mmˆ3] from baseline to days 14 and 28 | 14 and 28 days
Change in absolute neutrophil count [x10ˆ3/mmˆ3] from baseline to days 14 and 28 | 14 and 28 days
Change in absolute neutrophil count [/mmˆ3] from baseline to days 14 and 28 | 14 and 28 days
Change in absolute lymphocyte count [/mmˆ3] from baseline to days 14 and 28 | 14 and 28 days
Change in prothrombin time ratio from baseline to days 14 and 28 | 14 and 28 days
Change in partial thromboplastin time ratio from baseline to days 14 and 28 | 14 and 28 days
Change in bilirubin [mg/dl] from baseline to days 14 and 28 | 14 and 28 days
Change in lactate dehydrogenase [U/L] from baseline to days 14 and 28 | 14 and 28 days
Change in CPK-MB [ng/mL] from baseline to days 14 and 28 | 14 and 28 days
Change in troponin [ng/mL] from baseline to days 14 and 28 | 14 and 28 days
Change in von Willebrand factor antigen level (VWF:Ag) [%] from baseline to days 14 and 28 | 14 and 28 days
Change in von Willebrand factor activity (ristocetin cofactor) [%] from baseline to days 14 and 28 | 14 and 28 days
Change in ADAMTS-13 [%] from baseline to days 14 and 28 | 14 and 28 days
Change in von Willebrand multimeters from baseline to days 14 and 28 | 14 and 28 days
Change in plasminogen activator inhibitor-1 levels [ng/mL] from baseline to days 14 and 28 | 14 and 28 days
Change in E-selectin levels [ng/mL] from baseline to days 14 and 28 | 14 and 28 days
Change in P-selectin levels [ng/mL] from baseline to days 14 and 28 | 14 and 28 days
Change in endothelin [fmol/mL] from baseline to days 14 and 28 | 14 and 28 days
Change in circulating microparticles from baseline to days 14 and 28 | 14 and 28 days
Change in thromboelastography from baseline to days 14 and 28 | 14 and 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas, São Paulo, Brazil